CLINICAL TRIAL: NCT01014819
Title: A Phase I Clinical Trial of Dermacorder for Detecting Malignant Skin Lesions
Brief Title: A Clinical Trial of Dermacorder for Detecting Malignant Skin Lesions
Acronym: Dermacorder
Status: Completed | Type: Observational
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Ervin Epstein, MD Scientist, Children's Hospital & Research Center Oakland
Other Study IDs: 2009-36
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Basal Cell Carcinoma
Keywords: Dermacorder; Electric field; basal cell carcinoma; Gorlin Syndrome
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The Dermacorder measures the electric field in the skin. Malignant skin lesions disrupt the skin's normal electric field and this abnormal electric field can be detected by the Dermacorder. Therefore the investigators are testing the hypothesis that the Dermacorder can provide useful data to guide in the diagnosis of skin disease.

DETAILED DESCRIPTION:
The Dermacorder is a non-invasive medical device that scans a probe over the skin about 200 microns away from it and detects the electric field in the skin using capacitative coupling. Measurements of hundreds of malignant melanomas in mice indicated that these lesions generate an electric field that is easily detected. One previous clinical trial at the VA Medical Center in Hampton VA indicated an 80% reliability in predicting malignant lesions by their electric field. We have improved the Dermacorder over the past two years by enhancing its sensitivity and stability and must now determine if these improvements have improved its ability to detect malignant lesions. If the Dermacorder provides a reliable diagnosis of malignant lesions, its use could dramatically reduce the number of biopsies performed and this would significantly improve the quality of life for hundreds of thousands of Americans seeking the advice of dermatologists regarding suspicious lesions each year

ELIGIBILITY:
Inclusion Criteria:

* Study subjects must have had diagnosed at least one benign or malignant skin lesion;
* Subject is from 18-75 years of age, inclusive;
* Subject must sign and date all informed consent statements.

Exclusion Criteria:

* Subject is exhibiting signs of a bacterial or viral infection, including fever;
* Subject is unwilling to allow a biopsy of a malignant lesion for histological analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females with multiple basal cell carcinomas
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ervin Epstein, M.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Childrens Hospital Oakland Research Institute, Oakland, California, United States